CLINICAL TRIAL: NCT07109453
Title: Dermatological Safety Assessment of Test Products Using Primary Irritation Patch Test (PIPT) in Healthy Adult Human Subjects
Brief Title: To Assess Skin Safety of Test Product(s) by Patch Test on Adult Healthy Human Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Skin Harmony Lifescience Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB250037-SHL
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Normal; Sensitive Skin
MeSH Terms: interventions — Gene Expression

STUDY DESIGN:
Intervention Model Description: Primary Irritation Patch Test Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18 Test Products along with Positive and Negative Control (Experimental): 1. Deep Hydration Gel
  2. Anti-Wrinkle Gel
  3. Anti-Aging Gel
  4. Under Eye Cream
  5. Brightening Cream
  6. Moisturizing Cream
  7. Anti-Acne Serum
  8. Face Toner
  9. Anti-Aging Toner
  10. Clear Glow Toner
  11. Super Anti-Aging Serum
  12. Sun Screen SPF50
  13. Anti-Pigmentation Serum
  14. Super Cleansing Cream
  15. Root Revive Hair Serum
  16. Root Nourishment Hair Oil
  17. Anti-Acne Face Wash
  18. Ever Glow Face Wash 0.04 gm/ml of each Test Products along with positive control (1% SLS) and negative controls will be applied on the back of subjects i.e. between the scapula and waist through Finn chamber patch.
  Interventions: Other: 18 Test Products along with positive and negative control

INTERVENTIONS:
Other: 18 Test Products along with positive and negative control — 1. Deep Hydration Gel 2. Anti-Wrinkle Gel 3. Anti-Aging Gel 4. Under Eye Cream 5. Brightening Cream 6. Moisturizing Cream 7. Anti-Acne Serum 8. Face Toner 9. Anti-Aging Toner 10. Clear Glow Toner 11. Super Anti-Aging Serum 12. Sun Screen SPF50 13. Anti-Pigmentation Serum 14. Super Cleansing Cream 15. Root Revive Hair Serum 16. Root Nourishment Hair Oil 17. Anti-Acne Face Wash 18. Ever Glow Face Wash 0.04 gm/ml of each Test Products along with positive control (1% SLS) and negative controls will be applied on the back of subjects i.e. between the scapula and waist through Finn chamber patch.

SUMMARY:
To Check Dermatological Safety of Test Products by 24 Hours Patch Testing

DETAILED DESCRIPTION:
This is single center, evaluator-blinded study in healthy adult human subjects. Single 24-hour application of sponsor(s) provided test products along with positive and negative controls will be kept in contact with the skin of subjects under occlusion |Semi occlusion |Open patch for at least 24 hours (+ 2 hours). Study can be conducted in multiple groups. Safety will be assessed throughout the study by monitoring of adverse events. Subject's back i.e. between the scapula and waist will be utilized as application sites. Application sites will be evaluated for scoring the reaction, namely, erythema, dryness, and wrinkles on a 0-4 point scale separately for each parameter and oedema on another 0-4 points scale as per the Draize Scale after 30+5 minutes of patch removal, 24±2 hours and 168±2 hours after patch removal.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-65 years (both inclusive) at the time of consent.
* Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
* Subject with normal Fitzpatrick skin type III to V (Human skin colour determination scale).
* Females of childbearing potential must have a self-reported negative pregnancy test.
* Subject who do not have any previous
* history of adverse skin conditions and are not under any medication likely to interfere with the results.
* Subject is in good general health as determined by
* the Investigator on the basis of medical history.
* Subjects is willing to maintain the test patches in designated positions for 24 Hours.
* Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
* Subject must be able to understand and provide written informed consent to participate in the study.
* Subject is willing to refrain from vigorous physical exercise during the study period and follow all the instruction given.
* For Sensitive Skin Condition Only:
* Subject scoring greater than 30 for Section 2 - Sensitive v/s Resistant skin in modified Dr Baumann's* skin type questionnaire.
* Subject with sensitive skin as confirmed by Lactic Acid Stinging Test.

Exclusion Criteria:

* Subject having skin irritation, blemishes, excessive hair, moles, pigmentation, pimples, marks (e.g. tattoos (within the previous 3 months), scars, sunburn), open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the test site(s) i.e. back that can interfere with the reading.
* Medication which may affect skin response and/or past medical history.
* Subject having history of diabetes
* Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
* Subject suffering from any active clinically significant skin diseases which may contraindicate.
* Subject having history of any skin diseases including eczema, atopic dermatitis or active cancer.
* Participation in any patch test for irritation or sensitization within the last four weeks.
* Subject having history of asthma or COPD (Chronic obstructive pulmonary disease).
* Use of any:
* Prescribed or over-the-counter (OTC) anti-inflammatory drug within five (5) days prior to application.
* Antihistamine medication or immunosuppressive drugs within seven (7) days prior to first patch application. iii. Systemic or topical corticosteroids at patch site within four (4) weeks of test product application (steroidal nose drops and/or eye drops are permitted)
* Topical drugs used at application site.
* Subject with Self-reported Immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematous.
* Individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
* Subject with known allergy or sensitization to medical adhesives, bandages.
* Participation in other patch study simultaneously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the dermatological safety of the test products by 24 Hours Patch | Irritation Scoring at T30 minutes and 24 hours post patch removal. Scoring can be done at T168 hours post-patch removal if needed
  Test Dermatological safety of the test products by 24 Hours Patch Test will be evaluated by 0: No reaction and 4 Severe Reaction

SECONDARY OUTCOMES:
Safety of the skin | At T30 minutes and 24 hours post patch removal. Scoring can be done at T168 hours post-patch removal if required
  To evaluate the Safety of the skin by visual dermatological assessment by 0: No reaction and 4 Severe Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan Patel, Principal Investigator — NovoBliss Research Private Limited

IPD SHARING:
Plan to Share IPD: No